CLINICAL TRIAL: NCT06512207
Title: A Clinical Investigation on the Efficacy of Leuprorelin Acetate (Androgen Deprivation Therapy) Combined With Sintilimab (Anti-PD-1) in Advanced Lung Cancer
Brief Title: A Study on the Efficacy of Androgen Deprivation Therapy Combined With Anti-PD-1 Therapy in Advanced Lung Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jinzhou Medical University (Other)
Collaborators: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Yu Zhang, Professor, Jinzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NSFC-32230037
Record Dates: First submitted 2024-07-06; First posted 2024-07-22 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-08

CONDITIONS: NSCLC, Stage III; NSCLC, Stage IV
Keywords: Androgen Deprivation Therapy （ADT）; Leuprorelin acetate; NSCLC; PD-1 inhibitor
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Leuprolide; sintilimab; spartalizumab

STUDY DESIGN:
Intervention Model Description: 80 cases of stage III or IV NSCLC are randomly divided into two groups of 40 cases each. The control group is to receive conventional treatments (Chemotherapy + PD-1 Monoclonal Antibody), while the experimental group is to receive conventional treatments combined with Leuprorelin acetate.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional Treatment Group (Active Comparator): 40 cases in this group to receive the standard conventional treatment (Chemotherapy + PD-1 Monoclonal Antibody)
  Interventions: Drug: Sintilimab
- Conventional Treatment Combined with Leuprolide Group (Experimental): 40 cases in this group to receive the standard conventional therapy (Chemotherapy + PD-1 Monoclonal Antibody) combined with Leuprorelin acetate, 3.75 mg
  Interventions: Drug: Leuprorelin acetate + Sintilimab

INTERVENTIONS:
Drug: Leuprorelin acetate + Sintilimab — Leuprolide, an FDA-approved GnRH agonist, reduces sex hormone production and is widely used in clinical practice.
  Other Names: Leuprolide
  Arms: Conventional Treatment Combined with Leuprolide Group
Drug: Sintilimab — PD-1 inhibitor
  Other Names: Anti-PD-1 monoclonal
  Arms: Conventional Treatment Group

SUMMARY:
Androgen Deprivation Therapy (ADT) triggers thymic revitalization and increases thymic output, enhancing baseline anti-tumor immunity and responses to immunotherapies. Anti-tumor synergism has been identified by combining ADT with anti-PD-1 immunotherapy for androgen-independent tumors. This study is to investigate the combination of Leuprorelin ADT and Sintilimab (anti-PD-1) therapy in patients with advanced lung cancer.

DETAILED DESCRIPTION:
Immune checkpoint blockades (ICBs) are widely used in the clinical treatment of lung cancer. Studies have shown that the quantity and function of tumor-infiltrating lymphocytes (TILs) are associated with the effectiveness of PD-1 inhibitors in treating advanced NSCLC. The thymus is crucial for the differentiation, development, and maturation of T cells. With age, thymic atrophy leads to immunosenescence, significantly affecting baseline anti-tumor immunity and responses to immunotherapies. Preliminary findings have indicated that androgen deprivation therapy (ADT) not only directly induces apoptosis in prostate cancer cells but also may exert anti-tumor effects by promoting thymic regeneration. Furthermore, anti-tumor synergism has been identified by combining ADT with anti-PD-1 immunotherapy for androgen-independent tumors. Therefore, this study aims to investigate the combination of Leuprorelin ADT and Sintilimab (anti-PD-1) therapy in patients with advanced lung cancer.

ELIGIBILITY:
3.Inclusion Criteria:

1. Male patients aged ≥60 years.
2. ECOG performance status score of 0 ~1.
3. Expected survival time of more than 3 months.
4. Histologically or cytologically diagnosed advanced lung cancer according to the TNM staging system established by AJCC.
5. Patients who have not previously received any anti-PD-1 treatment.
6. Patients with adequate bone marrow function, no significant hepatic, renal, or coagulation dysfunction as per laboratory test criteria.
7. At least one tumor lesion meeting the following criteria:

   * No prior local treatments such as radiotherapy
   * Not biopsied during the screening period (if biopsy needed, baseline tumor assessment at least 14 days after the screening biopsy).
   * Measurable at baseline (longest diameter of the lesion ≥10 mm; For a lymph node, short diameter ≥15 mm).
   * If only one measurable lesion, no prior local treatments such as radiotherapy.
8. Ability to understand and voluntarily sign a written informed consent form.
9. Willingness to follow the study protocol and follow-up examinations.

Exclusion Criteria:

* Exclusion of cases that do not meet the inclusion criteria

Min Age: 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-12-03 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Complete Response (CR) | Efficacy evaluations are scheduled at 6 weeks,12 weeks and 18 weeks post treatment
  Disappearance of all target lesions, with nodular diseases excluded and target nodules reduced to <10mm in short axis.
Number of Participants with Partial Response (PR) | Efficacy evaluations are scheduled at 6 weeks,12 weeks and 18 weeks post treatment
  Reduction of at least 30% in the sum of diameters of all measurable target lesions compared to baseline
Number of Participants with Disease Progression (PD) | Efficacy evaluations are scheduled at 6 weeks,12 weeks and 18 weeks post treatment
  A 20% increase in the sum of the diameters of all measurable target lesions over the entire study period (using the smallest baseline value if it is the smallest), coupled with an absolute increase in the sum of diameters of at least 5mm. The appearance of one or more new lesions is also considered disease progression.
Number of Participants with Stable Disease (SD) | Efficacy evaluations are scheduled at 6 weeks,12 weeks and 18 weeks post treatment
  Lesion reduction not meeting PR criteria nor sufficient increase for PD, falling in between these two endpoints. The minimum sum of diameters during the study period can be used as a reference.
Quantity of Peripheral Blood Lymphocytes | Laboratory evaluations are scheduled before treatment, at 3 weeks post-treatment, and at 6 weeks post-treatment
  Assessment of peripheral blood lymphocyte quantity, comparing patients before and after a treatment cycle
Composition of Peripheral Blood Lymphocytes | Laboratory evaluations are scheduled before treatment, at 3 weeks post-treatment, and at 6 weeks post-treatment.
  Assessment of peripheral blood lymphocyte composition, comparing patients before and after a treatment cycle
Status of Recent Thymic Emigrants (RTEs) | Evaluations are scheduled before treatment, at 3 weeks post-treatment, and at 6 weeks post-treatment.
  Assessment of the status of Recent Thymic Emigrants (RTEs), comparing patients before and after a treatment cycle

CONTACTS AND LOCATIONS:
Overall Officials: Yu Zhang, Professor, Principal Investigator — Jinzhou Medical University
Locations (1):
- The Third Oncology Ward, First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No
We currently do not plan to share individual patient data (IPD) with other researchers due to confidentiality concerns and ethical restrictions. Additionally, the data collected in this study are considered proprietary and are crucial for ongoing and future research projects.